CLINICAL TRIAL: NCT04925791
Title: Does Limb Pre-Conditioning Reduce Pain After Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Michael Banffy, MD, Principal investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001182
Record Dates: First submitted 2021-06-09; First posted 2021-06-14 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hip Injuries; Hip Dislocation; Hip Fractures
MeSH Terms: conditions — Hip Injuries; Hip Dislocation; Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The IPC group (Experimental): subjects will get a standardized pre-conditioning treatment 24 hours prior to their hip arthroscopy. This consists of 3 rounds of 5 minutes of occlusion alternating with 5 minutes of reperfusion while seated.
  Interventions: Diagnostic Test: standardized pre-conditioning treatment
- The CON group (Other): subjects will get a controlled treatment of 20% of limb occlusion pressure 24 hours prior to their hip arthroscopy. This consists of 3 rounds of 5 minutes of minimal occlusion alternating with 5 minutes of reperfusion while seated.
  Interventions: Diagnostic Test: Partial occlusion

INTERVENTIONS:
Diagnostic Test: standardized pre-conditioning treatment — 3 rounds of 5 minutes of full occlusion alternating with 5 minutes of reperfusion while seated.
  Arms: The IPC group
Diagnostic Test: Partial occlusion — 3 rounds of 5 minutes of partial occlusion alternating with 5 minutes of reperfusion while seated.
  Arms: The CON group

SUMMARY:
The purpose of this study is to determine if the utilization of Ischemic Pre-Conditioning 24-hours prior to hip arthroscopy decreases patient's post-operative pain and opioid consumption.

DETAILED DESCRIPTION:
Subjects will be asked to take part in one of two treatment procedures 24 hours prior to their scheduled hip arthroscopy date. Subjects will be randomized into either the IPC or CON group.

These treatments consist of either 3 rounds of 5 minutes of occlusion alternating with 5 minutes of reperfusion or 3 rounds of 5 minutes of minimal occlusion alternating with 5 minutes of reperfusion. The treatment will last 30 minutes. Days 0-7 post-op will consist of self-reported pain scales and opioid consumption documentation in the morning and evening. This is a randomized single-blind research study.

This study has two study groups:

* The IPC group will get a standardized pre-conditioning treatment 24 hours prior to their hip arthroscopy. This consists of 3 rounds of 5 minutes of occlusion alternating with 5 minutes of reperfusion while seated.
* The CON group will get a controlled treatment of 20% of limb occlusion pressure 24 hours prior to their hip arthroscopy. This consists of 3 rounds of 5 minutes of minimal occlusion alternating with 5 minutes of reperfusion while seated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary hip arthroscopy by the PI between the ages of 18 and 55.

Exclusion Criteria:

* Patients younger than 18 or older than 55 who have had a previous hip arthroscopy, venous thromboembolism, and/or who take medications and/or supplements known to increase the risk of blood clots.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Pain levels VAS score | 7 days post op
  Pain score 0-10 with 0 being no pain and 10 being the worst

SECONDARY OUTCOMES:
number of days opioids were consumed post op | 7 days post op
  Total number days the patient had to take pain medication

CONTACTS AND LOCATIONS:
Overall Officials: Michael Banffy, MD, Principal Investigator — Cedar Sinai -Kerlan Jobe
Locations (1):
- Kerlan Jobe, Los Angeles, California, United States

REFERENCES:
- [Derived] Orner C, Usoro A, Bergeron B, Banffy M. Does Ischemic Preconditioning of the Operative Limb Reduce Pain After Hip Arthroscopy? A Prospective, Single-Blind, Randomized Controlled Trial. Orthop J Sports Med. 2025 Jun 10;13(6):23259671251343762. doi: 10.1177/23259671251343762. eCollection 2025 Jun. PMID 40502719